CLINICAL TRIAL: NCT00991887
Title: Radiation Therapy for Heterotopic Ossification Prophylaxis Acutely After Elbow Trauma
Acronym: ElbowHO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: there was an unacceptably high adverse event rate in the treatment group.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Orthopaedic Trauma Association (Other); OrthoCarolina Research Institute, Inc. (Other); Prisma Health-Upstate (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-04-09A
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2017-09

CONDITIONS: Elbow Fracture
Keywords: Heterotopic Ossification; Distal humerus Fracture-dislocations of the elbow; Radiation Therapy
MeSH Terms: conditions — Elbow Fractures; Ossification, Heterotopic | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Radiation Therapy (XRT) (No Intervention): This group will not receive radiation therapy after surgery.
- Radiation Therapy (XRT) (Active Comparator): Radiotherapy will be administered no later than 72 hours postoperatively.
  Interventions: Radiation: Radiation Therapy (XRT)

INTERVENTIONS:
Radiation: Radiation Therapy (XRT) — The dose will be 700 gray (derived unit of ionizing radiation dose in the International System of Units) in a single fraction, using AP-PA fields calculated to midplane. No Less than 6 MV energy photons will be used, and no bolus is placed on the skin. The field covers the entire joint, the antecubital fossa and the olecranon process. A strip of skin at the antecubital area is generally shielded, but is not an absolute requirement for this study.
  Other Names: Treatment group
  Arms: Radiation Therapy (XRT)

SUMMARY:
The investigators hypothesized that radiation therapy could be safely administered acutely after elbow trauma, and it would decrease the number of patients that would require surgical excision of heterotopic ossification.

DETAILED DESCRIPTION:
A multi-institutional, prospective randomized clinical trial will be employed to determine if single dose, limited field radiation therapy (XRT) will prevent post-traumatic heterotopic ossification (HO) after open reduction internal fixation of intra-articular distal humerus fractures and fracture-dislocations of the elbow and to assess function of the elbow after XRT and no XRT. Patients will be randomly assigned to one of the two groups(XRT/treatment or no XRT/control) by a computer-generated randomization schedule. Assignment will be in a ratio of 1:1 in a complete block design of 10. Each clinical site will be provided with a separate randomization assignment for each study participant. The treating surgeon and patient will be blinded to group assignment until after operative treatment. Clinical and radiographic assessments at 6 weeks, 3 months and 6 months post-operatively will be performed. The primary clinical outcome will be the Mayo elbow performance score which measures pain, stability, function and motion. Motion parameters (flexion, extension, pronation and supination) will be performed at each data collection point. Primary radiographic outcome will be the presence of heterotopic ossification by plain radiographs of the elbow in the antero-posterior and lateral planes at 6 weeks, 3 months, and 6 months post-operatively. Further imaging (radiograph or CT) will be obtained past the 6-month interval if deemed necessary by the treating physician,or if fracture union was not achieved at 6 months. The presence of HO will be quantified by radiograph. All adverse events will be documented. The trial will be monitored periodically by the Safety Monitor at least twice a year to ensure protocol compliance and address safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients with minimum age of 18 years and maximum age of 65.
* Patients deemed appropriate for operative intervention by the treating physician.
* Distal humerus intra-articular fractures (types 13-C1, C2, and C3), with or without proximal radius/ulna fractures - open or closed.
* Fracture-dislocations of the elbow (ulno-humeral dislocation associated with proximal ulna and/or radius fractures) - open or closed.

Exclusion Criteria:

* Head injury, quantified by Glasgow Coma Score (GCS) < 13 at time of consent for operative intervention.
* Burns > 20% Total Body Area (TBA) or involving the operative site.
* Patients with spinal cord injury affecting the upper extremities will be excluded.
* Open fractures which cannot be closed primarily within 72 hours of initial operative intervention.
* Patients with estimated life expectancy of less than one year due to preexisting condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-09; Primary Completion 2009-08 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bosse, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy (XRT): Radiotherapy will be administered no later than 72 hours postoperatively by a board-certified radiation oncologist. It was given as a single fraction at a dose of 700 cGy at 6-MeV energy photons with use of AP-PA (anteroposterior-posterioanterior) field calculated to midplane, with a mean window of 12x8.2cm, for all patients.
Period: Overall Study
Arm/Group | No Radiation Therapy (XRT) | Radiation Therapy (XRT)
Started | 26 | 22
Completed | 24 | 21
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Radiation Therapy (XRT) | Radiation Therapy (XRT) | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15) | 44 (17) | 45 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mayo Elbow Performance Score
Description: Mayo Elbow Performance Score (MEPS) is an outcome tool based on a 100 point scale, with higher score indicating better function. It measures pain, stability, function, and motion. The score is graded on the basis of the MEPS as excellent (>=90), good (75-89), fair (60-74), and poor (<60).
Time Frame: 6 month
Population: Patients with elbow trauma treated with radiation therapy in the prevention of post-traumatic heterotopic ossification. Subjects are randomized to either radiation therapy or no radiation therapy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Radiation Therapy (XRT) | Radiation Therapy (XRT)
Number analyzed (Participants) | 24 | 21
units on a scale | 66 (23) | 69 (19)

ADVERSE EVENTS:
Arm/Group | No Radiation Therapy (XRT) | Radiation Therapy (XRT)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 4/24 | 8/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Radiation Therapy (XRT) (N=24) | Radiation Therapy (XRT) (N=21)
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No